CLINICAL TRIAL: NCT02489708
Title: Pediatric Emergency Department Decision Support System to Reduce Secondhand Smoke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CINC 2014-5592; 1R21CA184337-01A1 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-07-03 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Asthma; Smoking Cessation
Keywords: Bronchiolitis; Cough; Ear Infection; Respiratory Infection; Wheezing; Clinical Decision Support Systems
MeSH Terms: conditions — Asthma; Smoking Cessation; Bronchiolitis; Cough; Otitis; Respiratory Tract Infections; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cessation Counseling (Experimental): Nurses will be trained to use Electronic Medical Record system to counsel families about second hand smoke exposure. Saliva samples will be obtained from 15 children at baseline and at follow-up to explore the effects of the nurse intervention.
  Interventions: Behavioral: Cessation Counseling

INTERVENTIONS:
Behavioral: Cessation Counseling — Nurses will be trained to use Electronic Medical Record system to counsel families about second hand smoke exposure. Saliva samples will be obtained from 15 children at baseline and at follow-up to explore the effects of the nurse intervention.

SUMMARY:
This two phase study will develop and evaluate a Pediatric Emergency Department (PED) Decision Support System (DSS)-Electronic Medical Records (EMR) System to facilitate the identification of smokers and the delivery of a Second Hand Smoke (SHSe) exposure intervention to caregivers who bring their child to the PED.

DETAILED DESCRIPTION:
The study will be the first to develop and evaluate a Pediatric Emergency Department (PED) Decision Support System (DSS)-Electronic Medical Records (EMR) System to facilitate the identification of smokers and the delivery of a Second Hand Smoke (SHSe) exposure intervention to caregivers who bring their child to the PED. The investigators will conduct a two-phased project to develop, refine, and integrate a Decision Support System into the current electronic medical record system. In Phase I, the investigators will develop a three-part DSS with prompts to: 1) ASK about child SHSe and caregiver smoking 2) Use a software program (REDCap) to ADVISE caregivers to reduce their child's SHSe via total smoking home and car bans and quitting smoking, and 3) ASSIST caregivers to quit by directly connecting them to their choice of free cessation resources (e.g., Quitline, txt2quit, smokefree.gov) during the PED visit. If the investigators discover that a teen participant is a smoker, the investigators will provide them with resources for the Quitline, tx2quit, and teen.smokefree.gov. The investigators will create reports to provide feedback to nurses on their SHSe counseling behaviors. Nurses will provide input on program content, functions, and design. In Phase II, the investigators will conduct a 3-month feasibility trial to test the results of implementing the DSS on changes in nurse SHSe-related behaviors, and child and caregiver outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who work at least 2 shifts per week
* Current smokers accompanying their 0-18 year old child to the Emergency Department or Urgent Care

Exclusion Criteria:

* Non English speaking families

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in Rate of Use of Decision Support System by Nurses | 3 months
Change in Amount of Second Hand Smoke Exposure in Children | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: E. Melinda Mahabee-Gittens, MD, MS, Principal Investigator — Professor
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Mahabee-Gittens EM, Dexheimer JW, Gordon JS. Development of a Tobacco Cessation Clinical Decision Support System for Pediatric Emergency Nurses. Comput Inform Nurs. 2016 Dec;34(12):560-569. doi: 10.1097/CIN.0000000000000267. PMID 27379524
- [Result] Mahabee-Gittens EM, Dexheimer JW, Khoury JC, Miller JA, Gordon JS. Development and Testing of a Computerized Decision Support System to Facilitate Brief Tobacco Cessation Treatment in the Pediatric Emergency Department: Proposal and Protocol. JMIR Res Protoc. 2016 Apr 20;5(2):e64. doi: 10.2196/resprot.4453. PMID 27098215
- [Derived] Mahabee-Gittens EM, Dexheimer JW, Tabangin M, Khoury JC, Merianos AL, Stone L, Meyers GT, Gordon JS. An Electronic Health Record-Based Strategy to Address Child Tobacco Smoke Exposure. Am J Prev Med. 2018 Jan;54(1):64-71. doi: 10.1016/j.amepre.2017.08.011. PMID 29102458